CLINICAL TRIAL: NCT01055795
Title: Phase I Study of the Combination of Bevacizumab, Everolimus and LBH589 (BEL) for the Treatment of Advanced Solid Tumors
Brief Title: Safety Study of Bevacizumab, Everolimus and LBH589 (BEL) for Advanced Solid Tumors
Acronym: BEL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herbert Hurwitz (Other)
Collaborators: Novartis (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Herbert Hurwitz, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00020190
Record Dates: First submitted 2010-01-24; First posted 2010-01-26 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Bevacizumab; Everolimus; Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab, Everolimus and LBH589 (Experimental): Dose Escalation Cohort #, Subjects, Bevacizumab, Everolimus, LBH589
  1. 3-6, All study drugs administered per dose level
  2. 3-6, All study drugs administered per dose level
  3. 3-6, All study drugs administered per dose level
  Expanded Cohorts Cohort #, Subjects, Bevacizumab, Everolimus, LBH589 A, B & C; 30, Recommended Phase II Dose for all three compounds
  Interventions: Drug: Bevacizumab, Everolimus and LBH589

INTERVENTIONS:
Drug: Bevacizumab, Everolimus and LBH589 — Dose Escalation Cohort #, Subjects, Bevacizumab, Everolimus, LBH589
  1. 3-6, All study drugs administered per dose level
  2. 3-6, All study drugs administered per dose level
  3. 3-6, All study drugs administered per dose level
  Expanded Cohorts Cohort #, Subjects, Bevacizumab, Everolimus, LBH589 A, B & C; 30, Recommended Phase II Dose for all three compounds

SUMMARY:
The main purpose of this study is to test the safety of three study drugs, bevacizumab (Avastin™), Everolimus (Afinitor™) and LBH589 (Panobinostat) when they are given together. It is hoped this study drug combination might lead to a greater decrease the in size of the cancer and/or slow down how fast the cancer is growing compared to when these drugs are given alone.

Subjects will be enrolled at Duke University Medical Center (DUMC).

DETAILED DESCRIPTION:
The main purpose of this study is to test the safety of three study drugs, bevacizumab (Avastin™), Everolimus (Afinitor™) and LBH589 (Panobinostat) when they are given together. It is hoped this study drug combination might lead to a greater decrease the in size of the cancer and/or slow down how fast the cancer is growing compared to when these drugs are given alone.

There are two parts of the study.

The purpose of part I is to find out the highest and safest levels of these drugs when they are given together. If you are enrolled in part I of the study, you will start all the study drugs at the same time. The amount (dose) of drugs you will get will depend on when you enter the study.

The purpose of part II is to see what effects, good and/or bad, the study drugs have when they are given alone and together. In addition, this will also give us a better understanding of how these study drugs work on you and your cancer. If you are enrolled in part II of the study, you will enter one of three study drug arms:

Study Drug Arm A: You will receive everolimus alone for two weeks, then add bevacizumab and LBH589 to your study regimen.

Study Drug Arm B: You will receive LBH589 alone for two weeks, then add bevacizumab and LBH589 to your study regimen.

Study Drug Arm C: You will receive everolimus and LBH589 together for two weeks, then add bevacizumab to your study regimen.

ABOUT THE STUDY DRUGS:

* Bevacizumab (Avastin™) is an intravenous (I.V., meaning through a vein) medication made from a special type of human and mouse protein called antibodies. Bevacizumab blocks a factor called VEGF (vascular endothelial growth factor) which is important for angiogenesis (the growth of new blood vessels). Blocking this factor is thought to block the growth of tumor-related blood vessels which may stop the growth of cancer. Bevacizumab and other drugs that block VEGF activity are currently being evaluated in clinical research studies in a variety of cancers.
* Everolimus (Afintor™) is a pill that works by blocking the activity of a substance in the body known as mTOR (mammalian target of rapamycin). mTOR is important for helping the growth and survival in normal and cancer cells. Blocking mTOR activity has been shown to slow or kill cancer cells in laboratory studies. Everolimus and other drugs that block mTOR activity are currently being evaluated in clinical research studies in a variety of cancers.
* LBH589 (Panobinostat) is a new pill that works by blocking a special group of proteins called histone deacetylases (HDACs). HDACs are important for helping the growth and survival in normal and cancer cells and for helping the growth of new tumor-related blood vessels. Blocking HDAC activity has been shown to shown to slow or kill cancer cells in laboratory studies. LBH589 and other drugs that block HDACs activity are currently being evaluated in clinical research studies in a variety of cancers. LBH589 (Panobinostat) is not approved by the U.S. Food and Drug Administration (FDA) for the treatment of cancer is therefore considered an investigational drug.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically confirmed malignant solid tumor that is refractory to standard therapies, or for which no standard therapies exist.
2. Patients must have at least one measurable site of disease according to RECIST (see Appendix 1) criteria that has not been previously irradiated. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation
3. Age ≥ 18 years
4. Karnofsky Performance status ≥ 80% (see Appendix 2)
5. Adequate bone marrow function as shown by:

   1. ANC ≥ 1.5 x 109/L
   2. Platelets ≥ 100 x 109/L
   3. Hemoglobin >9 g/dL; Erythropoietin and transfusion support is permitted provided treatments are not required more than every 8 weeks.
6. Adequate liver function as shown by:

   1. serum bilirubin ≤ 1.5 x ULN
   2. INR ≤ 1.5
   3. ALT and AST ≤ 2.5x ULN (≤ 5x ULN in patients with liver metastases)
7. Adequate renal function: creatinine clearance (estimated) ≥ 40 cc/min
8. Fasting serum cholesterol ≤ 300 mg/dL OR ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: Use of standard lipid lowering agents (see Section 10.3.6 for guidance) is permitted to meet eligibility.
9. Fasting blood sugar <160 mg/dL.
10. Baseline MUGA or ECHO must demonstrate LVEF ≥ 50%
11. TSH and free T4 within normal limits; Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism.
12. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days from day 1 of study drug and must be willing to use two methods of contraception, one of them being a barrier method during the study and for 3 months after last study drug administration
13. Signed informed consent

Exclusion Criteria:

1. Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks from day 1 of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.)
2. Patients who:

   1. have had a major surgery or significant traumatic injury within 4 weeks from day 1 of study drug,
   2. have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or
   3. are anticipated to require major surgery during the course of the study.
3. Patients with a known hypersensitivity to experimental drugs (or classes of drugs) or their excipients
4. Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent with the following exceptions:

   * Intermittent steroids ( not to exceed 4 mg every day) may be used on an as-needed basis (e.g. treatment for chemotherapy-related nausea.)
   * Patients on physiologic replacement doses of steroids due to adrenal insufficiency for any reason may remain on these medications.
   * Topical, inhaled or intra-articular corticosteroids
5. Patients should not receive immunization with attenuated live vaccines within one week of day 1 of study drug or during study period
6. Active brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases. Treated, asymptomatic metastases are permitted provided the patient has been off steroids for at least 1 month prior to day 1 of study drug.
7. Clinically significant arrhythmias including complete left bundle branch block or use of a permanent cardiac pacemaker, congenital long QT syndrome, history or presence of ventricular tachyarrhythmias, 2nd degree AV block type II, 3rd degree AV block clinically significant resting bradycardia (<50 beats per minute), QTcF > 450 msec on screening ECG.
8. Presence of poorly controlled atrial fibrillation (ventricular heart rate >100 bpm)
9. Previous history of CVA, TIA, angina pectoris, acute MI or history of recent re-perfusion procedures (e.g. PTCA) within 6 months from day 1 of study drug.
10. Congestive heart failure (New York Heart Association (NYHA classification, see Appendix 4 functional classification III-IV).
11. Fasting blood sugar > 160 mg/dL despite standard of supportive care. Patients may start or adjust anti-diabetic medications to meet eligibility.
12. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study as so judged by the treating physician. Examples include but are not limited to:

    1. Severely impaired lung function (e.g. use of home O2, history of Idiopathic Lung Disease (ILD), any evidence of ILD on scan.
    2. Active (acute or chronic) or uncontrolled severe infections requiring treatment with antibiotics
    3. Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
    4. Uncontrolled hypertension, BP>150/100 despite medical management
    5. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of oral medications (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
13. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to day 1 of study drug
14. History of hemoptysis (>/= 1/2 teaspoon of bright red blood per episode) within 1 month prior to day 1 of study drug
15. History of abdominal fistula or gastrointestinal perforation at any point within 6 months prior to day 1 of study drug, unless surgically repaired.
16. Use or need for full dose anticoagulation other than low molecular weight heparin (i.e. Lovenox only with and no other bleeding risk)..
17. Invasion or encasement of a major artery. Abutment without invasion or encasement is permitted. Abutment is defined as loss of the tissue plane between tumor and vessel but without invasion of the soft tissues or lumen of the vessel. Encasement is defined as more than 180 degrees of involvement
18. Serious, non-healing wound, active ulcer, or untreated bone fracture as judged by treating physician
19. Active, bleeding diathesis
20. Known history of HIV or Hepatitis B or C seropositivity
21. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. Two acceptable forms of contraceptives must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to day 1 of study drug)
22. Concomitant use of drugs with a risk of causing torsades de pointes (See Appendix 5 )
23. Concomitant use of CYP3A4 inhibitors (See Appendix 6)
24. Patients unwilling to or unable to comply with the protocol
25. Intrathoracic lung carcinoma of squamous cell histology. Mixed tumors will be categorized by the predominant cell type unless small cell elements are present, in which case the patient is ineligible; sputum cytology alone is acceptable. Patients with extrathoracic-only squamous cell NSCLC are eligible. Patients with only peripheral lung lesions (of any NSCLC histology) will also be eligible (a peripheral lesion is defined as a lesion in which the epicenter of the tumor is </= 2 cm from the costal or diaphragmatic pleura in a three-dimensional orientation based on each lobe of the lung and is </= 2 cm from the trachea, main, and lobar bronchi).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To define the maximal tolerated dose (if any) and the recommended phase II dose for the triplet combination of everolimus plus LBH589 plus bevacizumab in subjects with advanced solid tumors | 3 years

SECONDARY OUTCOMES:
To describe any dose limiting toxicities of this combination and to describe any non-dose limiting toxicities of this combination. | 3 years
To describe pharmacokinetic characteristics of everolimus and LBH589 when the two drugs administered in combination. | 3 years
To describe the effect of this treatment combination on blood based biomarkers for tumor angiogenesis and tumor growth factors. | 3 years
To describe any signs of clinical activity of this treatment combination, including response rate, time to progression, and duration of response. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Herbert I Hurwitz, Md, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States